CLINICAL TRIAL: NCT05517005
Title: An Exploratory Investigation of a B12 Vitamin to Increase Energy and Focus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sourse (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20248
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2022-08

CONDITIONS: B12 Deficiency Vitamin; Energy Supply; Deficiency; Mood
Keywords: Vitamin Deficiency; Energy; Mood-states; focus
MeSH Terms: conditions — Vitamin B 12 Deficiency; Avitaminosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hype Bites Supplement (Experimental): Participants will take the 2 chocolates each day, complete surveys at baseline, midpoint, and study conclusion, and take blood biomarker samples at baseline and conclusion
  Interventions: Dietary Supplement: Hype Bites Supplement

INTERVENTIONS:
Dietary Supplement: Hype Bites Supplement — The ingredients of the vitamin supplement are:
  Chocolate liquor Sugar Cocoa butter Vanilla extract Vitamin B12 (as methylcobalamin) Tapioca Gum arabic Coloring (radish, apple, black currant) Carnauba Wax

SUMMARY:
This study aims to examine the effects of Sourse's Hype Bites at being able to increase vitamin B12 levels to promote positive health outcomes. Participants will consume Hype Bites daily. Participants will also take surveys and blood samples to examine both the subjective experience of taking Hype Bites as well as changes in biomarkers across the trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 40 On a stable, consistent dietary regimen Must be on a vegan or vegetarian diet May experience the feeling of being tired often/several times a week. May experience brain fog May experience negative mood states

Exclusion Criteria:

* Females who are pregnant or breastfeeding Currently take vitamin B12 during the past four weeks Chronic conditions such has oncological of psychiatric disorders Anyone with IBS or IBD Anyone with a previous severe allergic reaction Anyone unwilling to follow the study protocol

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-05-22 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Examine if Hype Bites increase vitamin B12 in the blood | 8 weeks
  In order to examine the changes in B12, a blood sample will be used.

SECONDARY OUTCOMES:
examine the subjective improvements noticed by the study participants when supplementing with vitamin B12. | 8 weeks
  Questionnaires will be given to participants throughout the trial. These questionnaires will ask about changes in their ability to focus, concentrate, their energy levels, and their mood

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hill, PhD, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided